CLINICAL TRIAL: NCT01435876
Title: Treatment for Convergence Insufficiency Intermittent Exotropia; A Randomized Trial
Brief Title: Surgery and Convergence Insufficiency Intermittent Exotropia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sudhalkar Eye Hospital (Other)
Responsible Party: Principal Investigator, Aditya Sudhalkar, Dr. Aditya Sudhalkar, Sudhalkar Eye Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12132EH
Record Dates: First submitted 2011-09-13; First posted 2011-09-19 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Complications
MeSH Terms: interventions — Orthoptics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Surgical arm (Active Comparator): UNIOCULAR/BINOCULAR RECESSION/RESECTION PROCEDURES
  Interventions: Procedure: Post exercise Surgery
- Exercises (Active Comparator): ORTHOPTICS/MINUS LENS THERAPY
  Interventions: Procedure: Orthoptics
- Postoperative Exercises (Active Comparator): POST SURGICAL ORTHOPTICS/MINUS LENS
  Interventions: Procedure: Postop orthoptics
- Surgical (Active Comparator)
  Interventions: Procedure: Post exercises surgery

INTERVENTIONS:
Procedure: Post exercise Surgery — ORTHOPTICS/MINUS LENS THERAPY
  Other Names: Accomodative therapy
  Arms: Surgical arm
Procedure: Orthoptics — MINUS LENS THERAPY/ ORTHOPTICS
  Other Names: MINUS LENS THERAPY/ORTHOPTICS
  Arms: Exercises
Procedure: Postop orthoptics — ORTHOPTICS/MINUS LENS THERAPY
  Other Names: Minus Lens Therapy
  Arms: Postoperative Exercises
Procedure: Post exercises surgery — UNIOCULAR/BINOCULAR RECESSION/RESECTION
  Other Names: Minus Lens Therapy
  Arms: Surgical

SUMMARY:
This trial aims to determine which treatment modality is better for treatment of the convergence insufficiency subtype of intermittent exotropia.

DETAILED DESCRIPTION:
Surgery can give better results,

ELIGIBILITY:
Inclusion Criteria:Convergence Insufficiency Type Intermittent Exotropia

* No stereopsis
* Good visual acuity

Exclusion Criteria:

* Amblyopia
* Anisometropia > 2.5D
* Vertical deviations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2006-05; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Postoperative gain of stereopsis | 1month-1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aditya A Sudhalkar, M.S., Principal Investigator — Consultant
Locations (3):
- India (3):
  - Aditya Sudhalkar, Ahmedabad, Gujarat
  - M & J Institute Of Ophthalmology, Ahmedabad, Gujarat
  - M & J Institute, Ahmedabad, Gujarat